

## Cover Page Statistical Analysis Plan

Study Title: Modifying unconscious tongue movements to improve fluency in adults with a confirmed developmental stammer: a pilot randomized feasibility study

Document creation date: March 26th 2020

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]



Effect of treatment on primary outcome measure (percentage of participants with stammer <1.5% syllables) analysed by Chi square test and logistic regression analysis (ENTER method). The regression analysis to include the main effect of therapy, SSI-4 score, PAiS score where relevant and OASES-A. ANOVA will cater for type 1 error.